CLINICAL TRIAL: NCT03911193
Title: Phase II Single Arm Study With CABozantinib in Non-Small Cell Lung Cancer Patients With MET Deregulation
Brief Title: CABozantinib in Non-Small Cell Lung Cancer (NSCLC) Patients With MET Deregulation
Acronym: CABinMET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Ricerca Traslazionale (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABinMET
Record Dates: First submitted 2019-03-28; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cabozantinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): Elegible NSCLC patients with MET exon 14 skipping mutations or MET amplification will be treated with open label orally cabozantinib 60 mg/daily, cycles each 28 days.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Patients will be treated with cabozantinib 60 mg/daily (cycles each 28 days) until progression, toxicity or patient refusal.

SUMMARY:
This is a multicenter, single arm, phase II study evaluating efficacy in terms of RR in a cohort of NSCLC with MET amplification or MET exon 14 skipping mutation pre-treated or not with MET inhibitors.

DETAILED DESCRIPTION:
The study population will include NSCLC patients with MET amplification or MET exon 14 skipping mutation pre-treated or not with MET inhibitors. Elegible NSCLC patients with MET exon 14 skipping mutations or MET amplification will be treated with open label orally cabozantinib 60 mg/daily, cycles each 28 days. Disease evaluation will be performed every two months (8 weeks). Patients will be treated with cabozantinib until disease progression, unacceptable toxicity or patient refusal.Treatment will be continued until disease progression, unacceptable toxicity or patient refusal. Treatment beyond disease progression is allowed if considered appropriate by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Citological or histological diagnosis of non-small-cell-lung cancer (NSCLC) stage III B (not suitable for local treatments with curative intent) or stage IV.
2. Tissue samples available for MET analysis (archivial tissue or tissue collected at study entry); patients without archival tumor tissue or refusing new biopsy at study entry, are eligible if MET mutation is detected in cf-DNA
3. Presence of MET mutations (exon 14 skipping mutation ONLY) detected in tissue or cf-DNA at the local lab or in the central lab or MET amplification (MET/CEP7 ratio > 2.2) detected in the central lab ONLY.
4. Measurable disease according to RECIST criteria version 1.1
5. At least 1 prior line of standard therapy (chemotherapy and/ or immunotherapy)
6. Performance status 0-1 (ECOG)
7. Age ≥18 years
8. Patients potentially fertile using adequate methods of contraception in order to avoid childbearing. Contraceptive methods must be respected by male and female patients and their partners during study treatment period and at least 4 months after completing therapy
9. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to enrollment:

   1. ANC ≥ 1500 cells/μL without granulocyte colony-stimulating factor support
   2. Platelet count ≥ 100,000/μL without transfusion
   3. Hemoglobin ≥ 9.0 g/dL Patients may be transfused to meet this criterion
   4. AST, ALT, and alkaline phosphatase ≤ 2.5 × ULN, with the following exceptions:

      * Patients with documented liver metastases: AST and/or ALT ≤ 5 × ULN
      * Patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 × ULN.
   5. Serum bilirubin ≤ 1.25 × ULN
   6. Patients with known Gilbert disease who have serum bilirubin level ≤ 3 × ULN may be enrolled
   7. Calculated creatinine clearance (CRCL) ≥ 45 mL/min or calculated CRCL must be ≥ 60 mL/min
10. Patient compliance to the study procedure
11. Written informed consent

Exclusion Criteria:

1. Tissue sample not available in patients without MET exon 14 skipping mutation detected in cf-DNA
2. No possibility to assess MET status
3. Absence of any measurable disease according to RECIST criteria
4. Co-existence of driver events, including EGFR mutations, KRAS mutations, ALK rearrangements or ROS-1 rearrangements
5. No prior therapy
6. Concomitant chemotherapy or immunotherapy or radiotherapy
7. Symptomatic brain metastasis
8. Uncontrolled significant inter-current or recent illness, including cardio-vascular disorders and gastro-intestinal disorders
9. Major surgery within 2 months before first dose of study treatment
10. Concomitant anti-coagulation with oral anti-coagulants or plated inhibitors
11. History of significant bleeding, trachea-bronchial tree/major blood vessels invading tumors, cavity pulmonary lesions and GI disorders associated with a risk of perforation or fistula formation
12. Diagnosis of another cancer in the last 3 years, except for in situ carcinoma of cervix, breast and bladder or skin carcinoma (squamous or basalioid)
13. Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-09-21 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Response Rate (RR) (complete + partial responses) | Up to 36 months
  RR will be evaluated by investigators according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. Partial and complete responses will be confirmed following RECIST criteria 1.1. Disease evaluation will be performed every two months (8 weeks).

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 36 months
  Disease evaluation will be performed every 8 weeks
Overall survival (OS) | Up to 36 months
  Disease evaluation will be performed every 8 weeks
Disease Control Rate (DCR: stable disease + partial response + complete response) | Up to 36 months
  Disease evaluation will be performed every 8 weeks
Exploratory biomarkers | Up to 36 months
  At baseline, at the first disease evaluation and at progression of disease a blood sample will be collected for biomarkers analyses

CONTACTS AND LOCATIONS:
Overall Officials: Federico Cappuzzo, Principal Investigator — AUSL Romagna- P.O. di Ravenna
Locations (20):
- Italy (20):
  - A.O. "S.Giuseppe Moscati", Avellino, AV
  - IRCCS Oncologico Giovanni Paolo II, Bari, BA
  - A.O.U. Careggi, Florence, FI
  - Irccs Irst, Meldola, FO
  - Ospedale Infermi Rimini, Rimini, FO
  - A.O. Papardo, Messina, ME
  - Istituto Europeo di Oncologia, Milan, MI
  - Ospedale San Gerardo, Monza, MI
  - AOU Policlinico di Modena, Modena, MO
  - Casa di Cura La Maddalena, Palermo, PA
  - Istituto Oncologico Veneto, Padua, PD
  - A.O. S.M. Misericordia, Perugia, PG
  - Azienda Ospedaliero Universitaria Pisana, Pisa, PI
  - Azienda Ospedaliero- Universitaria di Parma, Parma, PR
  - AUSL Reggio Emilia- IRCCS Arcispedale S.M. Nuova, Reggio Emilia, RE
  - Fondazione Policlinico Gemelli, Roma, RM
  - Istituto Nazionale Tumori Regina Elena, Roma, RO
  - A.O.U. S. Luigi Gonzaga, Orbassano, Torino
  - AUSL della Romagna, Ravenna
  - Azienda Ospedaliero Universitaria Integrata di Verona, Verona